CLINICAL TRIAL: NCT05376150
Title: A Proof-of-Concept, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of XEN1101 in Major Depressive Disorder
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of XEN1101 in Major Depressive Disorder
Acronym: X-NOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-008-204
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Potassium channel; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- XEN1101 10 mg (Experimental): During the double blind treatment period (42 days), subjects will take 1 capsule of XEN1101 10 mg, orally with food, per day
  Interventions: Drug: XEN1101 10 mg
- XEN1101 20 mg (Experimental): During the double blind treatment period (42 days), subjects will take 1 capsule of XEN1101 20 mg, orally with food, per day
  Interventions: Drug: XEN1101 20 mg
- placebo (Placebo Comparator): During the double blind treatment period (42 days), subjects will take 1 capsule of placebo, orally with food, per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN1101 10 mg — XEN1101 oral capsule
  Arms: XEN1101 10 mg
Drug: XEN1101 20 mg — XEN1101 oral capsule
  Arms: XEN1101 20 mg
Drug: Placebo — Placebo capsule
  Arms: placebo

SUMMARY:
This is a multicenter, Phase 2, double-blind, randomized, parallel-arm, placebo-controlled clinical trial to evaluate the efficacy, safety, and tolerability of XEN1101 in subjects with Major Depressive Disorder.

DETAILED DESCRIPTION:
The study is divided into 3 stages: Screening - up to 4 weeks duration; Treatment - 6 weeks duration; Follow-up - 4 weeks duration. The total study duration per subject is estimated to be approximately 14 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Be properly informed of the nature and risks of the study and given written informed consent.
* Male or female, aged 18 through 65 years (inclusive) with a body mass index (BMI) ≤35 kg/m².
* Subject must meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for current MDD and currently in a moderate to severe major depressive episode (MDE), confirmed using the Mini International Neuropsychiatric Interview (MINI).
* Current MDE duration ≥2 months and <24 months at the time of screening.
* Current illness severity that is at least moderate, defined as a score of ≥20 on the HAM-D17 at screening and on Day 1.
* Score ≥20 on the SHAPS at screening and on Day1.
* Must be willing to comply with the study protocol for the full term of the study.

Key Exclusion Criteria:

* A primary psychiatric diagnosis other than MDD as defined by DSM-5 (comorbid anxiety disorders [including agoraphobia, generalized anxiety disorder, social anxiety disorder, post-traumatic stress disorder (PTSD), and panic disorder] are allowed).
* Concomitant use of antidepressants and/or other disallowed pharmacotherapy (including benzodiazepines).
* History of schizophrenia or other psychotic disorder, MDD with psychotic features, bipolar I or II disorder, or MDD with mixed features.
* History of non-response to >1 antidepressant drug due to lack of efficacy in the current MDE.
* Failing >3 antidepressant drug trials, for any reason, in the current MDE.
* History of non-response to electroconvulsive therapy (ECT) in the past 10 years.
* Active suicidal plan/intent in the past 6 months, or more than 1 lifetime suicide attempt.
* Females who are pregnant, breastfeeding, or planning to become pregnant during the first administration of study drug until 3 months after the last dose of study drug.
* Meets criteria for a substance use disorder within the past 12 months, with the exception of tobacco use, and/or has a positive urine toxicology screen for drugs of abuse.
* Any medical condition or personal circumstance that, in the opinion of the investigator, exposes the subject to unacceptable risk by participating in the study or prevents adherence to the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score. | From baseline to end of treatment (Week 6).
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From randomization to Week 10.

SECONDARY OUTCOMES:
Change in Snaith-Hamilton Pleasure Scale (SHAPS) score. | From baseline to end of treatment (Week 6).
Change in Beck Anxiety Inventory (BAI) score. | From baseline to end of treatment (Week 6).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (20):
- United States (20):
  - Advanced Research Center, Anaheim, California
  - Sunwise Clinical Research, LLC, Lafayette, California
  - California Neuropsychopharmacology Clinical Research Institute, Pico Rivera, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Meridian International Research, Miami, Florida
  - Global Medical Institutes (GMI), Miami, Florida
  - CCM Clinical Reseach Group, LLC, Miami, Florida
  - i-Research, Atlanta, Decatur, Georgia
  - Psych Atlanta, PC, Marietta, Georgia
  - iResearch, Savannah, Georgia
  - Revive Research Institute, Inc., Elgin, Illinois
  - Altea Research, Las Vegas, Nevada
  - Hassman Research Institute, Marlton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Neurobehavioral Research, Inc. (NBR), Cedarhurst, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Richard M Weisler and Association, Raleigh, North Carolina
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - AIM Trials, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butterfield NN, Luzon Rosenblut C, Fava M, Correll CU, Rothschild AJ, Murrough JW, Mathew SJ, Beatch GN, Grayson C, Harden C, Qian J, McIntosh J, Namdari R, Kenney C. Azetukalner, a Novel KV7 Potassium Channel Opener, in Adults With Major Depressive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2514278. doi: 10.1001/jamanetworkopen.2025.14278. PMID 40423966